CLINICAL TRIAL: NCT07069998
Title: Artificial Intelligent Guided Treatment of Atrial Fibrillation: A Randomized Controlled Pilot Study
Brief Title: AI-guided AF Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RD2025-05
Record Dates: First submitted 2025-05-21; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Placebo Comparator)
  Interventions: Other: Standard AF care
- Virtual Assistant (Experimental)
  Interventions: Other: virtual assistant

INTERVENTIONS:
Other: virtual assistant — Programming codes that interpret atrial fibrillation symptoms and design management plans based on algorithms that reflect the European Society of Cardiology (ESC) 2024 guidelines and the expertise of consultant cardiologists, finally checked and approved by a cardiologist.
  Arms: Virtual Assistant
Other: Standard AF care — AF care provided via the National Health System (NHS) standard AF care system
  Arms: Standard of Care

SUMMARY:
Two-centre, prospective, randomized, open-label, controlled pilot study to examine whether integrating an artificial intelligence virtual assistant (VA), instructed with the latest international guidelines on optimal patient management into the outpatient management of patients diagnosed with atrial fibrillation (AF) in the last 6 months, is feasible, acceptable and effective in reducing the need for regular medical assessment and the healthcare burden, reduce variability, and meets with participant satisfaction, without compromising participant safety and overall care quality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Documented diagnosis of AF within the last 6 months
3. Patient is at least mildly symptomatic. Presence of at least one of the symptoms like palpitation, dizziness, breathlessness, pre-syncope, and syncope with at least mild intensity
4. Ability to understand and comprehend the study rationale, design, and process.

Exclusion Criteria:

1. Severe comorbidities (such as physical impairment, cognitive impairment, and hearing loss) that could affect protocol adherence, in the opinion of the investigator
2. Chronic Kidney Disease (CKD) stage 4-5 or on dialysis
3. Medical illness with a life expectancy of less than 1 year
4. Alternative potentially reversible causes of AF (such as surgery, sepsis, or thyroid dysfunction)
5. Dementia or other cognitive impairment
6. Currently involved in another AF interventional clinical trial
7. Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2028-05-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
How acceptable is the Virtual Assistant (VA) system as assessed by Sekhon's Theoretical Framework of Acceptability (TFA) questionnaire. | 12 weeks
  The acceptability of the Virtual Assistant (VA) system will be assessed using an acceptability questionnaire adapted from the 2022 Sekhon et al. Theoretical Framework of Acceptability (TFA). The questionnaire will be completed separately by both patients and research administrators, with the resulting scores reflecting the overall acceptability of the intervention.
  The questionnaire employs Likert-type scales and includes the following TFA components, where the highest score shows greater acceptability in that component:
  Affective Attitude: 2 items (scored 0-10, where 0 = lowest acceptability and 10 = highest) Burden: 2 items (scored 0-10) Ethicality: 1 item (scored 0-5) Perceived Effectiveness: 1 item (scored 0-7) Intervention Coherence: 1 item (scored 0-5) Self-Efficacy: 2 items (scored 0-10) General Acceptability: 1 item (scored 0-5)
Patient-Reported Adherence to the Virtual Assistant (VA) System: 4-Item Feasibility Questionnaire | 12 weeks
  Adherence to the VA system, as a marker of feasibility, will be assessed using a 4-item questionnaire adapted from the study by An, M. et al. ("What really works in intervention? Using fidelity measures to support optimal outcomes." Physical Therapy, 100(5), pp. 757-765). This questionnaire will be completed by patients and is designed to evaluate key aspects of adherence.
  Each item is scored on a 4-point scale (0-3), with a total possible score of 12. Higher scores indicate greater adherence to the VA system.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] An M, Dusing SC, Harbourne RT, Sheridan SM; START-Play Consortium. What Really Works in Intervention? Using Fidelity Measures to Support Optimal Outcomes. Phys Ther. 2020 May 18;100(5):757-765. doi: 10.1093/ptj/pzaa006. PMID 31944249